CLINICAL TRIAL: NCT00429234
Title: Phase I Open-Labeled Trial of Gemcitabine and Dasatinib in Advanced Solid Tumors
Brief Title: Gemcitabine and Dasatinib in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0574
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Advanced Cancer; Solid Tumors
Keywords: Advanced Cancer; Solid Tumors; Dasatinib; BMS-354825; Sprycel; Gemcitabine; Gemcitabine Hydrochloride; Gemzar
MeSH Terms: interventions — Dasatinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib + Gemcitabine (Experimental): Dasatinib starting dose 70 mg by mouth daily for Week 1. Cycle is 28 days, except Cycle 1 which is 8 weeks. Gemcitabine starting dose of 800 mg/m^2 by vein once weekly over 30 minutes beginning Cycle 1 Day 1. All other cycles once weekly for 7 weeks on Days 8, 15, 22, 29, 36, and 43. Cycle is 28 days, except Cycle 1 which is 8 weeks.
  Interventions: Drug: Dasatinib; Drug: Gemcitabine

INTERVENTIONS:
Drug: Dasatinib — Starting dose 70 mg by mouth daily for Week 1. Cycle is 28 days, except Cycle 1 which is 8 weeks.
  Other Names: BMS-354825; Sprycel
Drug: Gemcitabine — Starting dose of 800 mg/m^2 by vein once weekly over 30 minutes beginning Cycle 1 Day 1. All other cycles once weekly for 7 weeks on Days 8, 15, 22, 29, 36, and 43. Cycle is 28 days, except Cycle 1 which is 8 weeks.
  Other Names: Gemzar; Gemcitabine Hydrochloride

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of dasatinib in combination with gemcitabine that can be given to patients with advanced solid tumors. The safety of this combination of study drugs will also be studied.

Researchers also want to study the pharmacodynamics (PDs) of this study drug combination. PD testing is used to learn what effect the drugs have on your tumors.

DETAILED DESCRIPTION:
Dasatinib is designed to block several proteins that have been shown to be important for the growth, spreading, and survival of cancers cells.

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause them to die and prevent further growth of cancer cells.

The amount of dasatinib and gemcitabine that you receive will depend on when you start on this study. There will be 3 participants enrolled in each group. The first group of participants enrolled on this study will be given small doses of dasatinib and gemcitabine. If no intolerable side effects are experienced, the next group of participants will be enrolled at a higher dose level. This process will continue until researchers find the highest tolerable dose of dasatinib and gemcitabine that can be given without intolerable side effects occurring. Up to 15 more patients will be enrolled at this highest tolerable dose in an expansion group. If you are enrolled in the expansion group, you will have a biopsy for PD testing prior to your first day on the study. Your doctor will tell you which group you are enrolled in.

Your study doctor will tell you what dose of dasatinib and gemcitabine you will be receiving and how it compares to the doses other participants have received. While on study, your dose may be increased to the next higher level, if the next higher dose level has already been tested in other participants and found to be tolerable.

You will take dasatinib by mouth once a day for 7 days in a row before you begin receiving gemcitabine by vein. If no intolerable side effects from dasatinib occur, you will continue taking it for the rest of the study. If you are enrolled in an expansion group, you will take dasatinib by mouth once a day for 56 days in a row.

If the disease get worse or you experience any intolerable side effects with dasatinib, you will be taken off this study before you begin taking gemcitabine.

You will receive gemcitabine by vein over 30 minutes starting on Day 8. The first cycle is 9 weeks long (63 days). You will receive gemcitabine by vein over 30 minutes once a week for 7 weeks on Days 8, 15, 22, 29, 36, 43, and 50. On Days 51-63, you will not receive any gemcitabine (a rest period for this drug), but you will continue to take dasatinib once a day. There will not be a rest period for dasatinib.

If you are enrolled in an expansion group, you will receive gemcitabine by vein over 30 minutes starting on Day 1. The first cycle is 8 weeks long (56 days). You will receive gemcitabine by vein over 30 minutes once a week for 7 weeks on Days 1, 8, 15, 22, 29, 36 and 43. On Days 44- 56, you will not receive any gemcitabine (a rest period for this drug), but you will continue to take dasatinib once a day. There will not be a rest period for dasatinib.

Cycle 2 and all other cycles will equal 28 days. You will continue to take dasatinib once a day. You will receive gemcitabine once a week for 3 weeks on Days 1, 8, and 15. On Days 16-28, you will not receive any gemcitabine, but you will continue to take dasatinib once a day.

If you experience any intolerable side effects, you may need to have additional blood drawn (about 2 teaspoons) to monitor your condition. Your dose level may be reduced to stop intolerable side effects from occurring, depending on what the study doctor thinks is best. If the disease gets worse or you continue to experience any intolerable side effects with gemcitabine, you will be taken off this study.

You will have blood drawn (about 1 teaspoon each time) for PD testing. In Cycle 1 before your daily dose of dasatinib and gemcitabine, PD blood samples will be drawn 1-4 days before you receive the study drug, on Day 8 (on the day the 1st dose of gemcitabine is given) and at the end of week 4 before your receive the study drug.

During Week 4 of Cycle 1 and at the end of Cycle 1, you will have a physical exam, including measurement of your vital signs. You will have blood drawn (about 1 tablespoon) and urine collected (at the end of Cycle 1 only) for routine tests. You will be asked how well you are able to perform the normal activities of daily living (a performance status evaluation) and how you are feeling. You will also be asked about other drugs you may be taking and if you have had any intolerable side effects from the study drugs.

On Day 1 of all remaining cycles, you will have a physical exam, including measurement of your vital signs. You will have blood drawn (about 1 teaspoon) for routine tests. You will have a performance status evaluation and be asked how you are feeling. You will also be asked about other drugs you may be taking and if you have had any intolerable side effects from the study drugs.

Once your participation has ended on this study for any reason, you will be asked to have an end-of-study visit that should occur about 28 days after the last dose of the study drug. At this visit, you will have a physical exam, including measurement of your vital signs and weight. You will have a performance status evaluation and be asked how you are feeling. Blood (about 1 teaspoon) and urine will be collected for routine tests. You will be asked about other drugs you may be taking, and you will be asked if you have had any intolerable side effects from the study drugs. Women who are able to have children will again have a blood (about 1 teaspoon) pregnancy test.

If there are study-related side effects reported at the end-of-study visit, you will continue to have follow-up visits or telephone calls, (which will last about 5-10 minutes each time) at least every 4 weeks, to check if you are still experiencing sides effects and until you no longer experience them.

This is an investigational study. Dasatinib and gemcitabine are both FDA approved and commercially available. Their use together in this study is experimental and authorized for use in research only. Up to 63 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Available for protocol-required follow-up
3. Eastern Cooperative Oncology Group (ECOG) performance status score 0 - 1
4. Histologic or cytologic diagnosis of a primary solid malignancy
5. Evidence (radiographic or tissue confirmation) that the disease is metastatic, or locally advanced in patients who are not candidates for standard therapy
6. Measurable disease, as defined by Response Evaluation Criteria In Solid Tumors (RECIST)
7. Adequate bone marrow function defined as: a) absolute neutrophil count (neutrophil and bands) >/= 1,500 cells/mm^3, b) platelet count >/= 100,000 cells/mm^3, c) hemoglobin >/= 9.0 g/dl
8. Adequate hepatic function defined as: a) total bilirubin </= 1.5 times the institutional upper limit upper limit of normal (ULN), b) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </= 2.0 times the institutional ULN, c) Exception: patients with primary liver tumors or known liver metastases: </= 3.0 times the institutional ULN for total bilirubin, AST and ALT
9. Adequate renal function defined as serum creatinine </= 1.5 times the institutional ULN
10. Serum potassium and magnesium levels within institutional normal limits. Total serum calcium or ionized calcium level must be greater than or equal to the lower limit of normal. Patients with low potassium, calcium and magnesium levels may be repleted to allow for protocol entry
11. Prior chemo-, radio-, hormonal or immunotherapy are allowed. Patients must have recovered from toxicity due to prior therapy i.e., toxicity has resolved to baseline or is deemed irreversible. At least 4 weeks must have elapsed since the last chemotherapy or investigational agent (6 weeks for nitrosoureas, mitomycin-C, and liposomal doxorubicin), immunotherapy or radiotherapy and the beginning of protocol therapy. At least 2 weeks must have elapsed since last hormonal therapy or exposure to any other "targeted" kinase inhibitor (e.g., imatinib mesylate)
12. Men and women, ages 18 and older
13. Women of childbearing potential (WOCBP) must be using an adequate method (i.e. barrier, spermicidal) of contraception to avoid pregnancy throughout the study and for a period of at least 1 month prior and at least 3 months after the study in such a manner that the risk of pregnancy is minimized
14. Continued from inclusion #13: WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea >/= 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL]
15. Continued from inclusion #13 and 14: Even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential
16. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication
17. At the MTD expansion phase of the protocol, all patients must have fine needle aspirate (FNA) biopsiable disease

Exclusion Criteria:

1. Women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method (i.e. barrier, or spermicidal) to avoid pregnancy for the entire study period including the period from one month prior to starting study medication and for a period of at least 3 months after the study
2. Women who are pregnant or breastfeeding
3. Women with a positive pregnancy test on enrollment or prior to study drug administration
4. Men who are unwilling or unable to use an acceptable method (i.e. barrier, or spermicidal) of birth control for the entire study period and for at least 3 months after completion of study medication if their sexual partners are WOCBP
5. Received extensive prior radiation therapy to the bone marrow. Generally, patients should have radiation to </= 25% of bone marrow-containing skeleton
6. Symptomatic brain metastasis that are either untreated or uncontrolled by surgery and or radiotherapy. Patients with symptoms of brain metastasis are not eligible unless brain metastasis are ruled out by CT or MRI and/or fully treated surgically or with whole-brain radiotherapy (WBRT)
7. A serious uncontrolled medical disorder or active infection which would impair the ability of the patient to receive protocol therapy
8. Uncontrolled or significant cardiovascular disease, including: a)A myocardial infarction within 6 months, b)Subjects with known symptomatic cardiomyopathy, c)Uncontrolled angina within 3 months, d)Congestive heart failure within 3 months, e)diagnosed or suspected congenital long QT syndrome, f)any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsade de pointes). Prolonged QTc interval on pre-entry electrocardiogram (>450 msec). If the automated reading is prolonged (i.e.>450 msec), the ECG should be manually overread,
9. Continued from exclusion #9: g) any history of second or third degree heart block (may be eligible if currently have a pacemaker) h) heart rate < 50 / minute on pre-entry electrocardiogram or i) uncontrolled hypertension
10. Dementia or altered mental status that would prohibit the understanding or rendering of informed consent
11. History of significant bleeding disorder including: a) Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease), b) Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies), c) Documented major bleeding episode from the GI tract within 6 months, d) Vasculitis, e) Evidence of organ dysfunction or digestive dysfunction that would prevent administration of study therapy
12. Patients who have not recovered from adverse events greater than grade 1 due to agents administered more than 4 weeks earlier
13. Prior exposure to dasatinib
14. Gastric pH modifying agents. Subjects should not take proton pump inhibitors and H2 antagonists. Short-acting antacid agents may be taken, and replaced for patients who are on gastric pH modifying agents prior to enrollment
15. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study
16. Because patients with immune deficiency are at increased risk of lethal infections when treated with myelosuppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with dasatinib or other agents administered during the study
17. Social situations that would limit compliance with study requirements
18. History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine, dasatinib, or other agents used in this study
19. Any pleural effusion felt to be clinically significant by the attending physician or principal investigator (P.I.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated combination doses (MTD) | 8 week cycle for Cycle 1, all other cycles 28 days

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org